CLINICAL TRIAL: NCT01185470
Title: THE CLINICAL EVALUATION OF IMPLANTABLE PUMP SYSTEM FOR SAFETY AND DELIVERY ACCURACY IN PATIENTS REQUIRING INTRATHECAL ADMINISTRATION OF MORPHINE SULFATE FOR CHRONIC PAIN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medallion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Cancers; Chronic Pain
Keywords: Chronic pain; Morphine Sufate; Intrathecal; Implantable drug delivery pumps
MeSH Terms: conditions — Neoplasms; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subjects with Implantable pump (Experimental): Patients with chronic pain responsive to intrathecal opioid analgesia as demonstrated in a morphine trial or patients with a previous successful intrathecal opioid therapy with an implantable pump will undergo study device implantation .
  Interventions: Device: Implantation of Morphine Sulfate delivering programmable pump

INTERVENTIONS:
Device: Implantation of Morphine Sulfate delivering programmable pump — Patients with chronic pain responsive to intrathecal opioid analgesia as demonstrated in a morphine trial or patients with a previous successful intrathecal opioid therapy with an implantable pump will undergo implantation of pump for intrathecal delivery of Morphine Sulfate.

SUMMARY:
• The objectives of this study are to confirm the medication delivery accuracy of the Infusion System, LLC Implantable Drug Delivery System (IDDS) with Patient Controlled Analgesia for intrathecal delivery of morphine sulfate for pain control, and to determine the safety profile of the system with PCA for intrathecal delivery of morphine sulfate for pain control.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 21 years of age.
2. Subject must have experienced chronic pain for at least 6 months.
3. Subject must not presently be on intrathecal therapy but must be considered a candidate for intrathecal analgesia by his pain specialist; or, a subject already on intrathecal therapy must be in need of a replacement intrathecal pump and catheter.
4. Subject must be capable of giving informed consent.
5. Subjects who agree to sign a Pain Treatment Agreement (Narcotic Contract) limiting narcotic prescriptions to the study physician.
6. Subjects who agree to periodic drug testing.
7. Subject must be capable and willing to follow all study-related procedures, including returning for monthly refills.
8. Subject must be cognitively intact and, in the opinion of the Investigator, capable of using the Patient Remote.
9. Subject who is not already successfully treated with intrathecal analgesic therapy must be responsive to a trial of intrathecal or epidural morphine.
10. Female subjects of child-bearing potential must agree to use a medically acceptable and effective double-barrier method of birth control.
11. Documented failure to respond to less invasive methods of pain control (such as physical or behavioral modifications).
12. Ineffective pain control with single or multiple systemic analgesic treatments (oral, rectal, IV or transdermal) or had intolerable side effects.
13. Cancer pain requiring strong opioids or non-malignant pain with average Visual Analog Scale (VAS) score of ≥ 4/10.
14. Subjects who can receive an MRI.
15. Subjects must be able to hear and respond to audible alarms or agree to have a support person available who is able to hear and respond to audible alarms.

Exclusion Criteria:

1. Subject is a female who is pregnant or is planning a pregnancy.
2. Subject is a nursing mother.
3. Subject has at the site chosen for implantation a skin condition that would prevent the implantation procedure.
4. Subject has participated in an investigational drug or device trial within 4 weeks prior to enrollment.
5. Subject has any known or suspected allergy to morphine or to the materials of the infusion pump or intrathecal catheter.
6. Subject shows signs of active, systemic infection.
7. Subject has a known central nervous system contraindication to intrathecal therapy, including but not limited to severe spinal canal stenosis or spinal cord compression.
8. Subject has a body size that is insufficient to accept the bulk and weight of the pump.
9. Subject is allergic to morphine sulfate, or for whom morphine sulfate is contraindicated.
10. Subject has a condition requiring diathermy procedures.
11. Subject has a life expectancy of less than 9 months.
12. Subject cannot independently comprehend and participate in the required assessments, including responding to the QOL, BPI, ODI and PGIC measurement tools.
13. Subject is not considered to be medically or psychologically appropriate for pump implantation.
14. Subject has a urine drug screen result which indicates the use of prescription drugs or controlled substances not on the order of a physician.
15. Subjects with an ASA Physical Status >IV.
16. Subjects with a history of spinal instability, or grade II spondylolisthesis or greater.
17. Previously implanted subjects with spinal MRI findings of inflammatory mass prior to the implantation procedures.
18. Subjects who are unable or unwilling to return to all of the required follow-up visits.
19. Subjects who are unwilling to sign the informed consent.
20. Subjects who are exposed to high-current industrial equipment (i.e. electricians or electrical engineers) or regularly exposed to MRI equipment (i.e. MRI technicians, MRI engineers and MRI clinicians).
21. Subjects with active implanted devices such as pacemakers, defibrillators, cochlear implants and neurostimulators or other medical device use that can interfere with the function of the implanted intrathecal pump.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
• Mean medication delivery accuracy. | 6 months
  Medication delivery accuracy will be evaluated at each of six (6) refills.

SECONDARY OUTCOMES:
• Tabulation of Adverse Events | 12 months
Concomitant Medications, Physical and Neurological Exam, Inflammatory Masses, Vital Signs, Incidence of Inflammatory Masses, Summary of COWS | 6 months
  Tabulation of Concomitant Medications, Tabulation of Physical and Neurological, Exam, Summary of Vital Signs, Incidence of Inflammatory Masses, Summary of COWS

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — The Center for Clinical Research
Locations (9):
- United States (9):
  - Center for Pain & Supportive Care, Scottsdale, Arizona
  - Coastal Pain Research, Carlsbad, California
  - University of California San Diego, La Jolla, California
  - Neurovations, Napa, California
  - Millenium Pain Center, Bloomington, Illinois
  - Global Scientific Innovations, LLC, Evansville, Indiana
  - Center for Pain Management, St Louis, Missouri
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Pain Research of Oregon, Eugene, Oregon